CLINICAL TRIAL: NCT06298682
Title: Characterization of Exosomes Platelets-released
Acronym: EXOPLT
Status: Recruiting | Type: Observational
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: CCM1421
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Platelet Thrombus
Keywords: exosomes, platelet activation, platelet inhibitors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — plasma, and platelets
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- subjects without known pathologies

SUMMARY:
Extracellular vesicles (EVs) play a key role in cell-to-cell communication. They are small vesicles that contain rich molecular cargo. Recently, they have been proposed as biomarkers for clinical diagnostics. EVs include three classes: small EVs (exosomes), large EVs (microparticles), and apoptotic bodies. Platelet-derived EVs (PEVs) are the most abundant class in human blood and can actively participate in numerous physiological and pathological processes. The information about the role of platelet exosomes in cardiovascular disease and the effect of antiplatelet agents on their release and content is very limited.

DETAILED DESCRIPTION:
This study is a multicentre, observational. We plan to enrol 54 subjects from Centro Cardiologico Monzino IRCCS, and 121 buffy coat related to 121 subjects from Centro Trasfusionale Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico. biographical and anthropomorphic data will be recorded, a fasting blood venous sample (from ante-cubital vein) will be collected for the haematochemical analyses and for research samples.

ELIGIBILITY:
Inclusion Criteria:

* subjects without known pathologies

Exclusion Criteria:

* individuals with gastrointestinal diseases,
* individuals with history of hepatic diseases,
* individuals with history of urogenital diseases,
* individuals with history of hematological diseases,
* individuals with history of immunological diseases,
* individuals with history of renal diseases,
* individuals with history of metabolic diseases
* individuals with history of respiratory diseases
* individuals with history of cancer
* individuals with history of cardiovascular disease
* individuals having permanent organ damage
* individuals with major trauma in the last 6 months prior to enrollment
* individuals with surgery in the last 6 months prior to enrollment
* individuals taking medication in the 15 days prior to enrolment.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: subjects without known pathologies
Sampling Method: Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2021-07-08 (Actual); Primary Completion 2026-07-07 (Estimated); Study Completion 2027-07-07 (Estimated)

PRIMARY OUTCOMES:
Characterization of exosomes released by activated platelet by Nanoparticle Tracking Analysis (NTA) and proteoma analysis | 36 month
Characterization of exosomes released by activated platelet and exposed to platelet inhibitors by NTA and proteoma analysis | 36 month

SECONDARY OUTCOMES:
Platelet exosome profile emerged by NTA and proteoma analysis will be related with the "biographical" and "anthropometric" data of the subjects. | 40 month

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy